CLINICAL TRIAL: NCT05969769
Title: Effects of Thoracic Manual Mobilization Techniques in Females of Coccydynia
Brief Title: Effect of Thoracic Mobilization in Females With Coccydynia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Laiba Zahid
Record Dates: First submitted 2023-07-23; First posted 2023-08-01 (Actual); Last update posted 2023-08-22 (Actual); Status verified 2023-08

CONDITIONS: Coccyx Disorder
Keywords: Coccyx Disorder; thoracic

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Active Comparator): Sustained Natural Apophyseal Glides will be performed with Muscle Energy Technique and Short Wave Diathermy as experimental group.
  Interventions: Other: Thoracic Sustained Natural Apophyseal Glides
- Control Group (Active Comparator): Short wave diathermy will be given with Muscle Energy Techniques.
  Interventions: Other: Muscle Energy Techniques

INTERVENTIONS:
Other: Thoracic Sustained Natural Apophyseal Glides — Sustained Natural Apophyseal Glides 3 sets of 10 reps with 1 min rest btw sets.
  Arms: Experimental Group
Other: Muscle Energy Techniques — Short wave diathermy for 10 to 15 mins Muscle Energy Techniques of following muscles will be performed, Hip flexors muscles, Quadrates lamborum muscles, Erector spinae muscles, Piriformis muscles, PFS technique of METs Isometric hold 5-7 sec, Stretching 15 sec, Rest 30 sec.
  Arms: Control Group

SUMMARY:
Coccydynia is common and prevalent among the females and several types of exercises and electrotherapy are advised. Pain can reduced significantly with both short wave diathermy and muscles stretches. There is limited evidence on indirect method like thoracic mobilization techniques to improve coccydynia. This study will determine the effects of thoracic mobilization techniques on coccydynia.

DETAILED DESCRIPTION:
Coccydynia, refers to pain in the coccyx region. it can be caused by various factor including trauma or injury (such as falls or child birth ), repetitive strain, prolong sitting on hard surface, or even idiopathic reasons. Treatment options for Coccydynia may include conservative measures, such as pain medication, using cushion or donut-shaped pillows to relieve pressure, applying heat or cold packs, and avoiding activities that's exacerbate the pain. Physical therapy including exercises such as stretching, Muscle Energy Technique (MET) can also be beneficial in some cases. Thoracic manual therapy, which involves hands-on techniques applied to the thoracic spine, can indeed be beneficial for improving spine mobility. While it may not directly target the coccyx itself, improving overall spinal mobility can have indirect effects on coccyx pain and dysfunction.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed females coccydynia patients.

Exclusion Criteria:

* Pregnancy
* 6 Months past Surgery, fracture or dislocation of coccyx.
* Malignancy or cyst in the pelvic area.

Ages: 20 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 44 (Estimated)
Dates: Start 2023-08-01 (Actual); Primary Completion 2024-01-01 (Estimated); Study Completion 2024-02-01 (Estimated)

PRIMARY OUTCOMES:
Numeric Pain Rating Scale | 8th Week
  Changes from the baseline Numeric Pain Rating Scale will be used to assess pain. • The Numeric Pain Rating Scale is an eleven-point measure of pain: the patient rates pain from 0 (no pain) to 10 (worst imaginable pain). The NPRS has shown good responsiveness in shoulder pain.
Modified OSWESTRY Low Back pain Index | 8th Week
  Changes from the baseline ODI is a disease specific disability measure is used to establish a level of disability stage on a patient activity status and monitor change over the time. The ODI is made up of 10 questions. Each question is scored from (o-5) m

CONTACTS AND LOCATIONS:
Overall Officials: summra andleeb, MS(OMPT), Principal Investigator — riphah internation university
Locations (1):
- Rahman Medical Hospital, Peshawar, KPK, Pakistan

IPD SHARING:
Plan to Share IPD: No